CLINICAL TRIAL: NCT02807207
Title: A Phase 1, Single-Center, Pacritinib- Versus Placebo-Blinded, Active- and Placebo-Controlled, Randomized, 3-Way Crossover Study to Evaluate the Cardiac Safety and Pharmacokinetics Following a Single Oral Dose Administration of Pacritinib in Healthy Subjects
Brief Title: To Evaluate the Cardiac Safety and PK Following a Single Oral Dose Administration of Pacritinib in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: PAC107
Record Dates: First submitted 2016-05-03; First posted 2016-06-21 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2016-06

CONDITIONS: Healthy Subjects
Keywords: To Study pharmacokinetics and Cardiac safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (6):
- Sequence I (Experimental): treatment sequence: A/B/C
  Interventions: Drug: A: pacritinib; Other: B: Placebo; Drug: C: moxifloxacin
- Sequence II (Experimental): treatment sequence: A/C/B
  Interventions: Drug: A: pacritinib; Other: B: Placebo; Drug: C: moxifloxacin
- Sequence III (Experimental): treatment sequence: B/A/C
  Interventions: Drug: A: pacritinib; Other: B: Placebo; Drug: C: moxifloxacin
- Sequence IV (Experimental): treatment sequence: B/C/A
  Interventions: Drug: A: pacritinib; Other: B: Placebo; Drug: C: moxifloxacin
- Sequence V (Experimental): treatment sequence: C/A/B
  Interventions: Drug: A: pacritinib; Other: B: Placebo; Drug: C: moxifloxacin
- Sequence VI (Experimental): treatment sequence: C/B/A
  Interventions: Drug: A: pacritinib; Other: B: Placebo; Drug: C: moxifloxacin

INTERVENTIONS:
Drug: A: pacritinib — Treatment A
  Other Names: A: pacritinib 400mg
Other: B: Placebo — Treatment B
Drug: C: moxifloxacin — Treatment C
  Other Names: C: moxifloxacin 400mg

SUMMARY:
The primary objective is to evaluate the cardiac safety of a single oral dose (400 mg) of pacritinib compared to placebo on the QT calculated using the Fridericia correction (QTcF) interval in healthy subjects.

DETAILED DESCRIPTION:
This is a randomized, pacritinib- versus placebo-blind, placebo- and active-controlled, single-dose, single-center, 3-period crossover study to evaluate the cardiac safety of a single 400-mg dose of pacritinib compared to placebo, and to characterize the PK of pacritinib and major human metabolites of pacritinib. The study is blinded for pacritinib and placebo, and open-label for moxifloxacin.

Subjects were to receive 3 treatments (400 mg pacritinib, placebo, and 400 mg moxifloxacin) in a crossover fashion. Each treatment is administered as monotherapy during 1 of 3 treatment periods with a 7-day washout period between administration of each study medication. Screening occurred up to 28 days before Check-in (Day -1) of Period 1. On Day -1 of Period 1, subjects checked into the Clinical Research Unit (CRU) for baseline assessments and were confined to the CRU for the remainder of the study until Study Completion (Day 22)/Early Termination. Continuous 12-lead cardiodynamic ECG monitoring and recording was performed from predose (at least

1 hour before administration of study medication) through 24 hours after the administration of study medication, then for 15 minutes every 12 hours (on Days 2 to 7 of each period). Blood samples for PK analysis were also collected predose (Hour 0) and at each cardiodynamic ECG timepoint postdose. Safety endpoints (eg, adverse events [AEs], clinical laboratory evaluations, vital signs) were monitored throughout each period. Subjects were discharged at Study Completion (Day 22). Subjects were scheduled to return for a Follow-up Visit 14 days (±3 days) later on Day 36.

ELIGIBILITY:
Inclusion Criteria:

1. healthy males or females, between 18 and 55 years of age, inclusive, who are non-tobacco users;
2. with BMI range from 18.0 to 32.0 kg/m2, inclusive;
3. normal or not clinically significant 12-lead ECG, in the opinion of the Investigator;
4. heart rate of 45 to 90 beats per minute (bpm), inclusive, after 5 minutes in the supine position;
5. mean systolic blood pressure <141 mmHg and mean diastolic blood pressure <90 mmHg, average value for each taken in duplicate at Screening (a repeat duplicate set may be performed once at Screening);
6. in good health, determined by no clinically significant findings from medical history, physical examination, and vital signs;
7. 7. clinical laboratory evaluations (including clinical chemistry panel [fasted at least 10 hours], CBC, and UA) within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator;
8. negative test for selected drugs of abuse (including alcohol) at Screening and at Check-in (Day -1 of Period 1);
9. negative hepatitis panel (including hepatitis B surface antigen [HBsAg] and hepatitis C virus antibody [anti-HCV]) and negative HIV antibody screens;
10. females must be non-pregnant and non-lactating, and females not of childbearing potential must be postmenopausal for at least 1 year or surgically sterile (eg, tubal ligation, hysterectomy) for at least 90 days, or agree to use, from the time of signing the informed consent or 10 days prior to Check-in (Day -1) of Period 1 until 30 days after Study Completion (Day 22)/ET, one of the following forms of contraception: non-hormonal intrauterine device (IUD) with spermicide; female condom with spermicide; contraceptive sponge with spermicide; intravaginal system (eg, NuvaRing®); diaphragm with spermicide; cervical cap with spermicide; male sexual partner who agrees to use a male condom with spermicide; sterile sexual partner; or abstinence. Oral, implantable, transdermal, or injectable contraceptives may not be used from the time of signing the informed consent or 10 days prior to Check-in (Day -1) of Period 1 until 14 days after the final dose administration. For all females, the pregnancy test result must be negative at Screening and Check-in (Day -1) of Period 1;
11. males will either be sterile or agree to use, from Check-in (Day -1) of Period 1 until 90 days following Study Completion (Day 22)/ET, one of the following approved methods of contraception: male condom with spermicide; sterile sexual partner; or use by female sexual partner of an IUD with spermicide; a female condom with spermicide; a contraceptive sponge with spermicide; an intravaginal system; a diaphragm with spermicide; a cervical cap with spermicide; or oral, implantable, transdermal, or injectable contraceptives. Subjects will refrain from sperm donation from Check-in (Day -1) of Period 1 until 90 days following Study Completion (Day 22)/ET;
12. able to comprehend and willing to sign an Informed Consent Form (ICF).

Exclusion Criteria:

1. presence of any of the following electrocardiographic abnormalities based on the safety ECG at Screening:

   1. QTcF interval >450 msec
   2. unusual T-wave morphology (such as bifid T-wave) or flattened low voltage T-waves
   3. PR interval >210 msec or <110 msec
   4. evidence of second- or third-degree atrioventricular block
   5. electrocardiographic evidence of complete left bundle branch block (LBBB), right bundle branch block, or incomplete LBBB or intraventricular conduction delay or QRS duration >110 msec;
2. history of syncope, cardiac arrest, cardiac arrhythmias, torsades de pointes, structural heart disease, a family history of long QT syndrome, or ongoing cardiac dysrhythmias of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) grade >3.0;
3. history or clinical manifestation of clinically significant cardiovascular, pulmonary, hepatic (eg, hepatitis), renal, hematologic, gastrointestinal (eg, celiac disease, peptic ulcer, gastroesophageal reflux, inflammatory bowel disease), metabolic, allergic, dermatological, neurological, or psychiatric disorder (as determined by the Investigator; appendectomy and cholecystectomy are not considered to be clinically significant disease);
4. significant abnormalities in liver function tests (any/all of alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase >1.5 x upper limit of normal [ULN]; gamma-glutamyl transferase >2 x ULN; or total bilirubin >1.3 x ULN), kidney function tests (serum creatinine > ULN), hypokalemia (defined as serum potassium <3.0 mEq/L) that is persistent and refractory to correction, or hypomagnesemia (defined as serum magnesium <1.4 mEq/L);
5. history of malignancy, except the following: cancers determined to be cured or in remission for ≥5 years, curatively resected basal cell or squamous cell skin cancers, cervical cancer in situ, or resected colonic polyps;
6. history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator;
7. history of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs except that appendectomy and hernia repair will be allowed;
8. history of Gilbert's Syndrome;
9. history or presence of an abnormal ECG, which, in the Investigator's opinion, is clinically significant;
10. history of alcoholism or drug addiction within 1 year prior to Check-in (Day -1) of Period 1;
11. use of tobacco- or nicotine-containing products within 6 months prior to Check-in (Day -1) of Period 1 and during the entire study;
12. consumption of alcohol- or caffeine-containing foods and beverages for 72 hours prior to Screening and during the entire study;
13. consumption of grapefruit-containing foods and beverages or other potent cytochrome P450 (CYP)3A4 inhibitors for 72 hours prior to Screening and during the entire study;
14. participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives or 30 days prior to Check-in (Day -1) of Period 1, whichever is longer, and during the entire study;
15. use of oral, implantable, injectable, or transdermal contraceptives within 10 days prior to Check-in (Day -1) of Period 1 or from the time of signing the informed consent (females only) until 14 days after the final dose administration;
16. use of any prescription medications and/or products within 14 days prior to Check-in (Day -1) of Period 1 and during the entire study;
17. use of any over-the-counter, non-prescription medications, vitamins, or minerals within 7 days prior to Check-in (Day -1) of Period 1 and during the entire study;
18. use of phytotherapeutic/herbal/plant-derived preparations within 7 days prior to Check-in (Day -1) of Period 1 and during the entire study;
19. poor peripheral venous access;
20. donation of blood from 30 days prior to Screening through Study Completion (Day 22)/ET, inclusive, or of plasma from 2 weeks prior to Screening through Study Completion (Day 22)/ET, inclusive;
21. receipt of blood products within 2 months prior to Check-in (Day -1) of Period 1;
22. any diarrhea or vomiting during the Screening period or at Check-in (Day -1) of Period 1;
23. any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
QT calculated using Fridericia correction (QTcF) interval | ECG: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  To evaluate the cardiac safety of a single oral dose (400 mg) of pacritinib compared to placebo

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  To characterize the pharmacokinetics of pacritinib, moxifloxacin, and major metabolites
Treatment emergent Adverse events | Day1 to Day 36
  To characterize the safety and tolerability of pacritinib following single dose administration in healthy subjects. The frequency of TEAEs is summarized by treatment, MedDRA (version 16.0) system organ class, and preferred term
time to Cmax (tmax) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  To characterize the pharmacokinetics of pacritinib, moxifloxacin, and major metabolites
area under the concentration-time curve (AUC) from Hour 0 to the last measurable concentration (AUC0-t) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  To characterize the pharmacokinetics of pacritinib, moxifloxacin, and major metabolites
AUC extrapolated to infinity (AUC0-∞) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  To characterize the pharmacokinetics of pacritinib, moxifloxacin, and major metabolites
Apparent terminal elimination rate constant (λz) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  To characterize the pharmacokinetics of pacritinib, moxifloxacin, and major metabolites
Apparent terminal elimination half-life (t1/2) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  To characterize the pharmacokinetics of pacritinib, moxifloxacin, and major metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Whitehurst, MD, Principal Investigator — Covance Clinical Research Unit
Locations (1):
- Covance Clinical Research Unit Inc., Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes